CLINICAL TRIAL: NCT06001671
Title: Antitumor Activity and Safety of BEBT-109, a Novel EGFR Inhibitor, in Previously Treated NSCLC With EGFR Exon 20 Insertion Mutations: a Phase 1B, Dose Escalation and Expansion Trial
Brief Title: Antitumor Activity and Safety of BEBT-109, a Novel EGFR Inhibitor, in Previously Treated NSCLC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Professor, Deputy Director of Thoracic Oncology Department, Hunan Province Tumor Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BEBT-109
Record Dates: First submitted 2023-08-07; First posted 2023-08-21 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: NSCLC

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BEBT-109 120mg (Experimental): BEBT-109 orally at an initial dose of 120 mg once daily.
  Interventions: Drug: BEBT-109
- BEBT-109 180mg (Experimental): BEBT-109 orally at an initial dose of 180 mg once daily.
  Interventions: Drug: BEBT-109
- BEBT-109 240mg (Experimental): BEBT-109 orally at an initial dose of 240mg (120mg bid) once daily.
  Interventions: Drug: BEBT-109

INTERVENTIONS:
Drug: BEBT-109 — BEBT-109 is based on the "3+3" model, with a dose ascent starting from 120mg qd

SUMMARY:
This clinical study was a first-in-human, phase 1B, single-center, single-arm, open-label, dose escalation and expansion trial that aimed to determine the safety, tolerability and efficacy of BEBT-109 in patients with locally advanced or metastatic NSCLC harboring EGFR exon20ins mutations who had received at least one line of previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Sign written informed consent before implementing any trial-related procedures;
* Age ≥18 years and no limit on the gender.
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC with EGFR exon20ins mutation according to assessments made in local laboratories.
* Previous treatment and type of mutation:

  1. Disease progression in doses extension cases may have been treated with an EGFR-TKI (e.g., gefitinib, erlotinib, eclitinib, afatinib, or dapatinib) and prior written test reports confirming EGFR T790M mutation.
  2. Disease progression after prior chemotherapy regimen and/or EGFR-TKI treatment in dose-extension cases, and prior written test reports confirming EGFR 20 exon insertion mutations.
  3. Disease progression following prior chemotherapy regimen and/or EGFR-TKI treatment in dose-extension cases, and prior written test reports confirming other rare mutations in EGFR (EGFR G719A, L861Q, or S768I point mutations).
  4. Patients who are intolerant to chemotherapy or EGFR-TKI and have no other effective treatment can also be admitted to the dose expansion group after judgment by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Patients with brain metastasis were only enrolled if the metastases were stable.
* Subjects had at least 1 measurable lesion that met the RECIST 1.1 criteria.
* If female subjects are of childbearing potential, adequate contraception (e.g., condoms, etc.) should be used, no breastfeeding should be used, and a negative pregnancy test before administration should be given.

Exclusion Criteria:

* Combined with any other malignancy (except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix).
* Genetic testing confirmed the presence of C-MET amplification, HER-2 amplification and KRAS mutations, and other genetic mutations that clearly confirm resistance to EGFR-TKI.
* From the last treatment of EGFR-TKI (such as erlotinib, gefitinib, eclitinib, afatinib or osimertinib, etc.) to the first administration of this clinical trial, the interval is less than 14 days or 5 half-lives (whichever is longer is the exclusion criterion), and the specific drugs involved are decided by the investigator based on comprehensive consideration.
* In the 4 weeks prior to the first administration of the study treatment, participants had used other anticancer drugs (including immune cell therapy) in the previous treatment regimen.
* Those who have not withdrawn from other clinical trials within 4 weeks prior to the first administration of the study treatment.
* Previous homogeneous drug restriction:

  1. Patients with EGFR mutation previously treated with osimertinib or other third-generation EGFR inhibitor drugs (eg, ivelitinib, emetinib, and eflotinib) ;
  2. EGFR exon20 insertion mutants have used drugs that target EGFR 20 exon insertion mutants (e.g. Poziotinib tarloxotinib TAK788 JNJ-61186372 CLN-081, etc.)
  3. Other EGFR rare mutations (EGFR G719A, L861Q, or S768I point mutations) have been treated with afatinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
DLT | 2 years
  Defined as one of adverse events defined by NCI CTCAE V5.0 from the first day to the 28th day of the treatment period.
MTD | 2 years
  If only 1 of 3 participants in a dose group has DLT, 3 additional subjects in this group will be tested at the same dose level; If no participants developed DLT, the next dose study was conducted; If 2 of the first 3 participants developed DLT or 2 of 6 participants developed DLT, the previous dose of the dose was the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
ORR | 2 years
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects
DCR | 2 years
  Defined as the proportion of subjects with complete remission (CR), partial remission (PR) and stable disease (SD) to the total subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China